CLINICAL TRIAL: NCT05744726
Title: Comparison of A-PRF vs Bone Wax in Hemostasis, Pain Relief and Healing Following Exodontia: A Single-blind Randomised Control Trial
Brief Title: Comparison of A-PRF vs Bone Wax in Hemostasis, Pain Relief and Healing Following Exodontia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Altamash Institute of Dental Medicine (Other)
Collaborators: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Rehan Ahmad, Demonstrator/Lecturer, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F.2-81/2022-GENL/338/JPMC
Record Dates: First submitted 2023-01-12; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Post-Extraction Socket Hemostasis; Post-Extraction Socket Pain Relief; Post-Extraction Socket Healing
Keywords: Platelet Rich Fibrin; Wound Healing; Tooth Extraction; Pain Severity; Bone wax
MeSH Terms: conditions — Pain | interventions — bone wax

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A-PRF (Experimental): Advance Platelet-Rich Fibrin
  Interventions: Biological: A-PRF
- Bone-wax (Active Comparator)
  Interventions: Combination Product: Bone-wax
- Conventional Dental Extraction protocol (No Intervention): Control Group

INTERVENTIONS:
Biological: A-PRF — 0.5 to 1g of Advance Platelet-Rich Fibrin (A-PRF) clot for each dental socket.
  Arms: A-PRF
Combination Product: Bone-wax — 0.5 to 1g of Bone-wax for each dental socket
  Other Names: combination of beeswax and other products
  Arms: Bone-wax

SUMMARY:
The goal of this clinical trial is to compare the pain relief and healing effect of A-PRF and Bone-wax in patients having mandibular tooth-extractions. The main question[s] it aims to answer are:

In the perspective of improvement in pain and healing;

* Does A-PRF performs better than control group?
* Does Bone-wax performs better than control group?
* Healing index and Pain scale score Comparison of A-PRF and Bone-wax; if one is better than the other? Participants will be asked to give resoponse to a post-operative symptom severiety (PoSSe) scale. An investigator will score the patient's extraction for hemostasis and on healing index [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items]. If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects].

ELIGIBILITY:
Inclusion Criteria:

* All patients who need extraction of mandibular posterior teeth
* Overall, systemically healthy individuals (Established based on history, i.e., patients who do not take medicine for any systemic condition).
* INR within normal range.

Exclusion Criteria:

* Patients with a diagnosed systemic condition.
* Patients who are immunocompromised.
* Patients who are unwilling to participate or withdraw from the study.
* Patients who fail to report on the seventh and twenty-first post-extraction day.
* Patients with physical or mental impairments who need assistance in taking their medications.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain Relief on VAS | 21 days
  Patients receiving any of the intervention will be evaluated at just before, 3rd, 7th and 21st day of dental extraction on Visual Analogue Scale (VAS).
Extraction socket healing | 21 days
  Patients receiving any of the intervention will be evaluated at 3rd, 7th and 21st day of dental extraction on Healing index by Landry et al.

SECONDARY OUTCOMES:
Hemostasis | 30 minutes
  The post-operative bleeding will be evaluated 30 minutes after the placement of the last suture as:
  * No bleeding
  * Mild Bleeding: bleeding that stopped spontaneously or with minimal local compression.
  * Severe Bleeding: bleeding that did not stop with the previous measures and that required local adrenaline or continuous local compression using gauze pack soaked in the corresponding antifibrinolytic agent until the bleeding stops

CONTACTS AND LOCATIONS:
Locations (1):
- Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
As per institutional data privacy policy we are bound of not sharing patient data with other researchers

REFERENCES:
- [Background] Ruta DA, Bissias E, Ogston S, Ogden GR. Assessing health outcomes after extraction of third molars: the postoperative symptom severity (PoSSe) scale. Br J Oral Maxillofac Surg. 2000 Oct;38(5):480-7. doi: 10.1054/bjom.2000.0339. PMID 11010778
- [Background] Landry RG, Turnbell RS, Howley T (1988) Effectiveness of benzydamine HCL in treatment of periodontal post-surgical patients. Res Clin Forums 10:105-118.
- [Background] Yelamali T, Saikrishna D. Role of platelet rich fibrin and platelet rich plasma in wound healing of extracted third molar sockets: a comparative study. J Maxillofac Oral Surg. 2015 Jun;14(2):410-6. doi: 10.1007/s12663-014-0638-4. Epub 2014 Jun 28. PMID 26028867